CLINICAL TRIAL: NCT02894905
Title: An Open-label, Single-dose Study to Evaluate the Effect of Renal Impairment on the Single-dose Pharmacokinetics of AL-335
Brief Title: A Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of AL-335
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108225; 64294178HPC1009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — adafosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AL-335 (Cohort 1) (Experimental): Participants with mild impaired renal function will receive a single oral dose of AL-335 800 milligram (mg) (given as 2*400-mg tablets).
  Interventions: Drug: AL-335
- AL-335 (Cohort 2) (Experimental): Participants with moderate impaired renal function will receive a single oral dose of AL-335 800 mg (given as 2*400-mg tablets).
  Interventions: Drug: AL-335
- AL-335 (Cohort 3) (Experimental): Participants with severe impaired renal function will receive a single oral dose of AL-335 800 mg (given as 2*400-mg tablets).
  Interventions: Drug: AL-335
- AL-335 (Cohort 4) (Experimental): Participants with normal renal function will receive a single oral dose of AL-335 800 mg (given as 2*400-mg tablets).
  Interventions: Drug: AL-335

INTERVENTIONS:
Drug: AL-335 — Participants with various degrees of impaired renal function (mild [Cohort 1], moderate [Cohort 2], severe [Cohort 3]) and normal renal function (Cohort 4) will receive a single oral dose of AL-335 800 mg (given as 2*400-mg tablets).

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of a single oral dose of AL-335 in participants with various degrees of impaired renal function (mild, moderate, and severe) compared to participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1-4:

* Participant must have a body mass index (BMI; weight in kilogram (kg) divided by the square of height in meters) of 18 to 36 kilogram per meter square (kg/m^2), extremes included, and a body weight not less than 50.0 kg
* Participants must agree to follow all requirements that must be met during the study as noted in the Inclusion and Exclusion Criteria (eg, contraceptive requirements)
* Female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 30 days after study drug administration
* Male participant must agree not to donate sperm from enrollment (Day 1) in the study until at least 30 days after receiving the study drug

Cohorts 1-3:

* Participant must have stable renal function
* Participant must be otherwise healthy except for the renal impairment and its underlying disease states and mild comorbidities and participant must be medically stable on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening
* Participants must have an estimated glomerular filtration rate (eGFR) less than (<) 90 milliLiter per minute per 1.73 meter square (mL/min/1.73m^2). Mild renal impairment (eGFR 60 to <90 mL/min/1.73m^2); moderate renal impairment (eGFR 30 to <60 mL/min/1.73m^2); severe renal impairment (eGFR <30 mL/min/1.73m^2 not requiring dialysis)

Cohort 4:

* Participant must be healthy on the basis of physical examination, medical history, vital signs, 12-lead ECG, and clinical laboratory tests performed at screening
* Participants must have an eGFR greater than or equal to (>=) 90 mL/min/1.73m^2

Exclusion Criteria:

Cohorts 1-4:

* Participant has a history of any illness (unrelated to renal impairment or its underlying disease, as appropriate) that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant. This may include but is not limited to history of relevant drug or food allergies, history of cardiovascular or central nervous system disease, history or presence of clinically significant pathology, chronic skin disease, or history of mental disease
* Participant who is on a vegetarian diet or who takes creatine supplements, and who has a non-standard muscle mass, example (eg), amputation, malnutrition, muscle wasting, or extremely muscular (body building)
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening
* Participant who smokes more than 10 cigarettes or 2 cigars or 2 pipes per day from within 3 months before screening until the end of the study
* Participant is a woman who is pregnant, or breast-feeding, or planning to become pregnant from signing of the Informed Consent Form (ICF) onwards until 30 days after study drug administration
* Participant is a man who plans to father a child while enrolled in this study (Day 1) until 30 days after study drug administration.

Cohorts 1-3:

* Participant requires dialysis
* Participant with imminent renal replacement therapy (ie, during the study period)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of AL-335 | Pre-dose, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 28, 32, 36, 48, 60, and 72 hours post-dose
  The Cmax is the maximum observed concentration of analyte (AL-335).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Pre-dose, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 28, 32, 36, 48, 60, and 72 hours post-dose
  The AUClast is the area under the analyte (AL-335) concentration-time curve from time zero (0) to time of the last quantifiable concentration.
Area Under the Concentration-Time Curve From Time Zero to Infinite Time (AUCinfinity) | Pre-dose, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 28, 32, 36, 48, 60, and 72 hours post-dose
  The AUCinfinity is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to follow-up (Approximately 30-35 days after study drug administration)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Orlando, Florida
  - Knoxville, Tennessee